CLINICAL TRIAL: NCT05383846
Title: Exposing Narrative Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 21041
Record Dates: First submitted 2022-04-25; First posted 2022-05-20 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2022-05

CONDITIONS: Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: Naturalistic, mixed-method, explanatory sequential measurement single case series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Narrative Exposure Therapy (Experimental): This is a multiple baseline single case series design which focuses on assessing the posited exposure and autobiographical memory integration components of Narrative Exposure Therapy; no comparator will be included.
  Interventions: Other: Experimental Narrative Exposure Therapy

INTERVENTIONS:
Other: Experimental Narrative Exposure Therapy — NET (Schauer et al., 2011) is an evidence-based, short-term, manualised treatment for complex trauma, aiming to reduce symptoms of traumatic stress in individuals. NET combines principles of CBT, Testimony Therapy, and Exposure Therapy.
  This is a multiple baseline single case series design which focuses on assessing the posited exposure and autobiographical memory integration components of Narrative Exposure Therapy; no comparator will be included.

SUMMARY:
The main purpose of the study is to further develop an existing measure of autobiographical memory integration (ABMI) to investigate and clarify the ABMI change process specific to narrative exposure therapy (NET).

DETAILED DESCRIPTION:
Traumas are events which include witnessing or being at the risk of, death, violence, and sexual violation. Experiencing trauma can lead to psychological and physiological changes, and an individual's mental health can deteriorate to the point where a diagnosis of Post-traumatic stress disorder (PTSD) is given; 10-20% of people develop enduring symptoms, with effective treatment being a challenge.

While being exposed to trauma does not lead to PTSD, there is a dose-response relationship between the severity and duration of traumatic events and developing PTSD, suggesting that more complex forms of PTSD can develop if a person is subjected to multiple traumatic events. Complex post-traumatic stress disorder (CPTSD) occurs when a person is subjected to multiple prolonged traumas of an interpersonal nature, where escape is impossible. Different treatment approaches are needed for PTSD and CPTSD.

One therapy which has received support for treating CPTSD is Narrative Exposure Therapy (NET). NET is a National Institute for Health and Care Excellence recommended short-term manualised therapy. NET appears to be a well-tolerated treatment and has consistently low attrition rates when compared to other therapies. There is also emerging evidence of NET's effectiveness in the general population. The central aim of NET treatment is re-integration of contextual information and the traumatic memory into an autobiographical lifeline; this occurs through narrating the memory and involves prolonged exposure and habituation, and integration of the trauma memory into an autobiographical context. Despite NET's successes, its mechanisms of change have not been evidenced empirically, especially the element of contextualisation and integration of trauma into autobiographical memory (ABM). Four participants will be recruited with the support of local staff working in mental health services across Nottinghamshire. Participants will receive between twelve to fourteen weekly interventions sessions. Changes will be explored through process and outcome measures administered before, during, and after the intervention and interviews will be conducted at the end to gather participants experiences.

The study is supported by The University of Nottingham. Potential benefits include providing participants with an intervention to resolve their trauma and also to provide a theoretical contribution by either proving or refuting the process measures posted by NET.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-65
2. Are able to give fully informed consent
3. Experiencing traumatic stress resulting from multiple traumatic events (no formal diagnosis of PTSD/CPTSD is needed)
4. Are able to communicate verbally and are fluent in English
5. Have no on-going current trauma focused therapy
6. Appropriate and ready for NET
7. Referred to either Step 4 Psychological Services or Centre for Trauma

Exclusion Criteria:

1. Under the age of 18.
2. Above the age of 65.
3. Currently experiencing an episode of psychosis.
4. Have an intellectual disability.
5. Are actively suicidal.
6. Are non-fluent in English.
7. Are currently abusing substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in autobiographical memory integration during NET intervention. A coding manual has been created by the research team to assess the posited mechanism of change- Autobiographical Memory Integration Coding Tool | Throughout intervention phase of the study, for approximately 24-28 weeks
  A coding manual has been created by the research team to assess the posited mechanism of change.
  The primary outcome (process) measure is autobiographical memory integration (ABMI) as this is a posited mechanism of change in NET. An existing coding measure (Jager et al., 2014; Lane, 2019) has been adapted for the purpose of the study, to include more areas measuring phenomenological constructs of autobiographical memory. The coding measure that has been created by the researcher will cover areas such as: Total word count of narratives (Gray & Lombardo, 2001); disorganisation (Harvey & Bryant, 1999)- repetition of phrases, confusion, and disjointedness; fragmentation (Foa et al., 1995)- unfinished thoughts, repetition of words, speech filler; vividness; time and place details; emotional distancing and sensory details (Boyacioglu & Akfirat, 2014). The measure will be used to code transcripts on a session-by-session basis and is therefore a process measure (primary aim of study).

SECONDARY OUTCOMES:
Change in symptoms of post-traumatic stress disorder between the baseline, NET intervention, and up to 1 month follow-up phase- as assessed by the Impact of Events Scale Revised (IES-R; Weiss & Marmar, 1997) | Throughout the study, for approximately 32 weeks ]
  The IES-R (Weiss & Marmar, 1997) will be used every session to assess symptoms of post-traumatic stress disorder. It is a 22 item self-report questionnaire, and is divided into three subscales, with 8 items on intrusion and avoidance: 6 on hyperarousal. The measure assesses Intrusion, avoidance and hyperarousal in PTSD over the last seven days. Answers on the measure ranges from 0 = Not at all; 1 = A little bit; 2 = Moderately; 3 = Quite a bit; 4 = Extremely, there are no specific cut off scores; however, scores over 24 indicate concern, with higher scores related to higher levels of distress.
Change in depression, anxiety, and stress between the baseline, NET intervention, and up to 1 month follow-up phase- as assessed by the Depression Anxiety and Stress Scale 21 (DAAS-21; Lovibond & Lovibond, 1995) | Throughout the study, for approximately 32 weeks
  The DAAS-21 (Lovibond & Lovibond, 1995) will be used every session to assess depression, anxiety, and stress, it is a self-report questionnaire ranging over the last seven days. The DAAS-21 measures general psychological distress as an outcome measure (secondary aim of study). The measure consists of 21 items which are divided into 3 subscales with 7 questions for each subscale. Answers range on a scale from 0= Did not apply to me at all; 1= Applied to me to some degree, or some of the time; 2= Applied to me to a considerable degree or a good part of time; 3= Applied to me very much or most of the time. Scores of 10 and above on the depression sub scale indicates mild difficulties with depression; 8 and above on the anxiety sub-scale indicates mild difficulties with anxiety, and 15 and above on the stress sub-scale indicates mild difficulties with stress.
Changes in heart rate and heart rate variability during the NET intervention, as assessed by the Polar H10 chest strap | Throughout the intervention phase of the study, for approximately 24-28 weeks
  The Polar H10 chest strap will be used to collect heart rate data (heart rate- HR and heart rate variability- HRV). The Polar H10 has been shown to be a reliable and valid measure of HR and HRV; even when compared to an ECG as gold standard (Gilgen-Ammann et al., 2019; Speer et al., 2020). HRV measures physiological arousal and is the variation in time between heartbeats, by taking 5-minute segments of heart rate recordings, will allow for visual analysis of the root mean square of the successive differences between R-R intervals (rMSSD). HRV will be Measured every session pre- and post-narration and re-narration and used as a before and after measure to see how it changes over therapy.
Process measure of habituation: Subjective Unit of Distress (SUD; Wolpe, 1969) | Throughout the intervention phase of the study, for approximately 24-28 weeks
  The process of exposure and habituation are typically measured through Subjective Units of Distress Scale (SUDS; Foa & Kozack, 1986; Wolpe & Lazarus, 1966), which is a person's subjective account of distress on a set scale. Participants will be asked to rate their level of distress on a scale from 0 (no distress) to 10 (maximum distress), at the start, middle, and end of their trauma narrations. This is to see if how this relates to HR data.
Change in body awareness and autonomic reactivity during NET session, as assessed by the Body Perception Questionnaire Short Form - Autonomic Nervous System (Porges, 1993, 2015) | Throughout the intervention phase of the study, for approximately 24-28 weeks ]
  The Body Perception Questionnaire Short Form (BPQ-SF; Porges, 1993; Kolacz et al., 2018) is a 46 item self-report measure that assesses a person's perception of body awareness and autonomic reactivity. The measure's items are based on the autonomic nervous system, and a set of neural pathways that connect the brain and body. It assesses a person's experiences of reactivity in their organs and tissues that are regulated by the autonomic nervous system. . The first domain and subscale is body awareness with high scores reflecting hypersensitivity, whereas low scores reflect low hyposensitivity. The second domain, Autonomic Reactivity has two subscales, Supradiaphragmatic Reactivity which measures the responses of autonomically-innervated organs above the diaphragm. The second subscale Subdiaphragmatic Reactivity measures the response of autonomically-innervated gastrointestinal organs below the diaphragm.

OTHER OUTCOMES:
Change Interviews (Elliot et al., 2001) | At 1 month follow up
  The feasibility and acceptability of the study will be investigated by conducting follow up change interviews with participants approximately one month after completing the treatment. In this instance, the participant will be asked to provide feedback on their experience of receiving treatment, including in terms of barriers and fascinators to engagement. The interviews will be conducted by an external researcher, i.e. another Trainee Clinical Psychologist. The interviews will be recorded and sent to the researcher and they will then be transcribed, after transcription content analysis will be applied to them.
Number of Traumatic Events- The Life Events Checklist (Weathers et al., 2013). | 1 week at consent session
  The Life Events Checklist (LEC-5) which is part of the PCL-5 will be used in the proposed study. The LEC-5 is not an outcome measure but will be used to assess the number and type of traumatic events a person has experienced which is being collected as demographic information.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sabin-Farrell, PhD, Principal Investigator — University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No